CLINICAL TRIAL: NCT01932307
Title: Cervical Spine Health of Surgeons
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H13-01151
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Occupational Health Physicians; Neck Pain
Keywords: Surgeon neck health
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PGY1 General Surgery Residents (Experimental): All first year general surgery residents at the University of British Columbia
  Interventions: Procedure: Neck strengthening exercise program

INTERVENTIONS:
Procedure: Neck strengthening exercise program — Study subjects will be introduced to a 2-minute neck strengthening exercise program and advised to follow for 10 weeks. The exercise program will include five different exercises that will strengthen the neck and stabilize the scapula. The exercises are: Chin retraction, cracking the egg, scapular clock, wall pushup and scapula retraction. Each will be completed as 3 isometric holds, 3 repetitions per set and 2 sets per exercise.

SUMMARY:
There are currently no standardized programs addressing the well-documented neck pain in surgeons as a result of non-ergonomic positioning and the use of microsurgical equipment. The primary goal of this study is to introduce a brief neck strengthening exercise program to optimize surgeons' neck health. Instructional videos outlining the program along with surveys designed to assess attitude towards neck health will be distributed to first year general surgery residents at the University of British Columbia (UBC) through their required online curriculum webpage. A followup survey will be administered 10 weeks later to determine efficacy of the program through self-reported adherence and changes in attitude towards neck health.

DETAILED DESCRIPTION:
1. Purpose:

   To evaluate the efficacy of a pre-operative 2-minute exercise program in reducing surgical residents self-reported neck pain.
2. Hypothesis:

   A 10 week 2-minute neck strengthening exercise program completed between cases will reduce self-reported chronic neck pain caused by the use of surgical instruments and increase musculoskeletal health awareness in a group of residents.
3. Justification:

   Surgical residents will be asked to complete a baseline survey regarding their self-rated neck pain. Then they will be introduced to a 2-minute neck strengthening exercise to be performed in between surgical cases. They will be asked to evaluate their neck pain again 10 weeks later.

   Neck pain experience before and after the introduction of neck exercises will be compared.
4. Objectives:

   1. Define the problem through prevalence data in a sample of surgeons.
   2. Understand qualitatively and quantitatively measures of pain and quality on residents.
   3. Evaluate the efficacy of a pre-operative 2-minute exercise program.
   4. Disseminate our results and change the cultural norms of practice.
5. Research Method:

   All first year general surgery residents at the University of British Columbia will be invited to participate. They will be asked to complete a survey regarding neck pain experience and introduced to a 2-minute neck muscle exercise video which they will be advised to follow for the next 10 weeks. Another follow-up survey will be sent at the end of 10 weeks.
6. Statistical analysis:

Percentage of residents showing >50% improvement using an alpha of 0.05 statistical significance will be the primary outcome measure using the appropriate validated pain questionnaire. The attitude of the residents towards their neck health before the intervention will be compared to their attitudes at the completion of the study using a Pearson's chi squared test as a measure of significant difference. The self-reported effectiveness and adherence of the program at the completion of the study will be used as a measure of efficacy. All statistical analysis will be conducted in SAS 9.3.

ELIGIBILITY:
Inclusion Criteria:

* All first year general surgery residents at the University of British Columbia

Exclusion Criteria:

* Previous serious neck injury (e.g. herniated disc)
* Chest pain during physical exercise
* Heart failure
* Spinal Stenosis
* Radicular nerve pain
* Neurological condition causing chronic pain
* Currently involved directly with the study group

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Neck pain and quality of life questionnaires | 10 weeks
  The subjects will be asked to complete the Bournemouth Neck Disability index online once at the start of the study and again following a 10 week period where the subjects will be encouraged to follow our exercise routine in between surgical cases.

SECONDARY OUTCOMES:
Adherence and attitudes towards the exercise program | 10 weeks
  A followup survey will be distributed 10 weeks following the exposure to the exercise program to determine self-reported adherence and attitudes to the program.

CONTACTS AND LOCATIONS:
Overall Officials: York NH Hsiang, MB MHSc FRCSC, Principal Investigator — Professor of Surgery, Division of Vascular Surgery, Department of Surgery
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada